CLINICAL TRIAL: NCT01679184
Title: XM-One Study for Living Donor Program
Status: Terminated | Type: Observational
Why Stopped: Lack of staff to enroll patients in this study
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Giselle Guerra, Assistant Professor of Clinical, University of Miami
Other Study IDs: XM-One
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Transplant; Failure, Kidney

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A total of 6 teaspoons of blood will be drawn.
Oversight: Data Monitoring Committee: No

SUMMARY:
Donor-Specific Antibody (DSA) (HLA) levels and non-HLA antibody levels in recipients prior to living kidney transplantation and randomize these individuals into a desensitization protocol in order to evaluate shifts that can occur with the Luminex and XM-One assay after treatment and up to 6 months post transplant.

If desensitization is needed prior to transplantation in individuals with a negative crossmatch but positive DSA and/or XM-one - patients will be evaluated clinically with routine lab tests (serum creatinine levels, spot urine protein and spot urine creatinine levels) as well as protocol biopsy evaluations.

DETAILED DESCRIPTION:
1. Rates of acute rejection including subclinical rejection - acute T cell mediated (cellular) rejection, antibody mediated acute rejection, and chronic antibody-associated injury (i.e.: Transplant Glomerulopathy, Chronic allograft arteriopathy) between the groups.
2. Evaluation of endothelial cell activation and injury on biopsies by checking markers for endothelial cell activation and injury (intercellular adhesion molecule-1, ICAM-1/CD54; vascular cell adhesion molecule-1, VCAM-1/CD106; and E-selectin, ELAM-1/CD62E) in two-color stains of tissue with classical endothelial markers (CD34 and Factor VIII).
3. Measurement of serum/plasma levels of TNF-alpha and VEGF and decreased levels of protein C and protein S in the circulation, as an assessment of graft vascular perturbation.
4. Circulating Endothelial Cells (CECs) will be measured by flow cytometry with markers for endothelial cell activation.

ELIGIBILITY:
Inclusion Criteria:

* Recipients receiving deceased donor transplants.
* Living donor transplant that is T-cell flow crossmatch positive.
* HIV, Hepatitis C and B positive patients.

Exclusion Criteria:

* Pregnant women and children will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living donor kidney transplant recipients
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
DSA | 1 year
  To evaluate Donor-Specific Antibody (DSA) (HLA) levels with Luminex testing and non-HLA antibody levels using XM-One assay in recipients before and after transplantation for up to 6 months as well as in those recipients undergoing desensitization treatment.

SECONDARY OUTCOMES:
DSA | 1 year
  Rates of acute rejection including subclinical rejection - acute T cell mediated (cellular) rejection, antibody mediated acute rejection, and chronic antibody-associated injury (i.e.: Transplant Glomerulopathy, Chronic allograft arteriopathy) between the groups.
  Determine role of desensitization prior to transplantation in individuals with a negative crossmatch but positive DSA and/or XM-one - based on Luminex and XM-One testing. Patients will be evaluated clinically with routine lab tests (serum creatinine levels, spot urine protein and spot urine creatinine levels) as well as protocol biopsy evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Guerra, R.N., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States